CLINICAL TRIAL: NCT02125201
Title: Effectiveness of Intranasal Versus Intravenous Fentanyl in Preterm and Term Newborns for Pain Prevention
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Peniakov Marina, Doctor, HaEmek Medical Center, Israel
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EMC-0089-13 - CTIL
Record Dates: First submitted 2014-03-21; First posted 2014-04-29 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Pain
Keywords: intranasal fentanyl; newborn
MeSH Terms: conditions — Pain | interventions — Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- intranasal fentanyl (Experimental): Intranasal Fentanyl 1.5-2 mcg/kg
  Interventions: Drug: Fentanyl
- intravenous fentanyl (Active Comparator): Intravenous Fentanyl 1-1.5 mcg/kg
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Fentanyl — A neonate will recieve Fentanyl intranasal or intravenous 5 minutes before the procedure The nurse will check his pain scale If the pain scale will be more than 4 the neonate will recieve the second dose of Fentanyl
  Other Names: Beatryl

SUMMARY:
Neonatal intensive care unit patients undergoes many painful procedures during their hospitalization. Effective pain control in such procedures as intubation, catheterization, central line insertion, chest tube insertion, etc. is an important part of treatment. Opioids administration is a common practice for acute pain prevention. Fentanyl is the preferred opioid due to it rapid onset and short duration of action.

Fentanyl may be given intravenously, transcutaneous transmucosal and intranasal. Intranasal administration is practiced for about 20 years. A rich vascular supply in a nose provides rapid absorption of the drug. This uninvasive root is now popular for pain prevention and treatment. There are about 20 trials with intranasal fentanyl administration to children from 6 month old to 18 years. The investigators did not find information about this way of administration in neonates.

In our pilot study the investigators want to check if intranasal administration of fentanyl is safe and effective in pain prevention in term and preterm neonates during invasive procedures and to compare it with intravenous route of administration.

ELIGIBILITY:
Inclusion Criteria:

Term and preterm neonates that require invasive procedures (elective or semielective intubation, central line insertion , chest drain or abdominal drain)

Exclusion Criteria:

1. Neonates with prolonged analgesic treatment before the procedure
2. Neonates with neurologic problem which can interact with pain assessment

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2014-06; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Pain scale - N-PASS | before the intervention and till one our after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Marina Peniakov, MD, Principal Investigator — HaEmek Medical Center, Israel
Locations (1):
- NICU, Afula, Israel